CLINICAL TRIAL: NCT02953587
Title: Effect of Ghrelin on Glucose Metabolism After Bariatric Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Naji Abumrad, John L. Sawyers Professor of Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 111237-Protocol II; R01DK091748 (NIH)
Record Dates: First submitted 2016-09-22; First posted 2016-11-03 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity | interventions — Glucose Tolerance Test; Ghrelin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vertical Sleeve Gastrectomy (VSG) NJ/PO (Experimental): Patients that are undergoing routine VSG will be studied preoperatively, and at 1 month postoperatively. Each time point will have two study visits with a cross-over design. The first visit at each time point will be randomized to a human ghrelin or a saline infusion, with the alternate infusion at the second visit. At each study visit, an Oral Glucose Tolerance Test (OGTT) will be performed by administering glucose through a nasojejunal (NJ) feeding tube preoperatively and orally (PO) postoperatively.
  Interventions: Procedure: Oral Glucose Tolerance Test (OGTT); Drug: Human Ghrelin; Drug: Saline
- Roux-en-Y Gastric Bypass (RYGB) NJ/PO (Experimental): Patients that are undergoing routine RYGB will be studied preoperatively, and at 1 month postoperatively. Each time point will have two study visits with a cross-over design. The first visit at each time point will be randomized to a human ghrelin or a saline infusion, with the alternate infusion at the second visit. At each study visit, an Oral Glucose Tolerance Test (OGTT) will be performed by administering glucose through a nasojejunal (NJ) feeding tube preoperatively and orally (PO) postoperatively.
  Interventions: Procedure: Oral Glucose Tolerance Test (OGTT); Drug: Human Ghrelin; Drug: Saline
- Vertical Sleeve Gastrectomy (VSG) PO/PO (Experimental): Patients that are undergoing routine VSG will be studied preoperatively, and at 1 month postoperatively. Each time point will have two study visits with a cross-over design. The first visit at each time point will be randomized to a human ghrelin or a saline infusion, with the alternate infusion at the second visit. At each study visit, an Oral Glucose Tolerance Test (OGTT) will be performed.
  Interventions: Procedure: Oral Glucose Tolerance Test (OGTT); Drug: Human Ghrelin; Drug: Saline
- Roux-en-Y Gastric Bypass (RYGB) PO/PO (Experimental): Patients that are undergoing routine RYGB will be studied preoperatively, and at 1 month postoperatively. Each time point will have two study visits with a cross-over design. The first visit at each time point will be randomized to a human ghrelin or a saline infusion, with the alternate infusion at the second visit. At each study visit, an Oral Glucose Tolerance Test (OGTT) will be performed.
  Interventions: Procedure: Oral Glucose Tolerance Test (OGTT); Drug: Human Ghrelin; Drug: Saline

INTERVENTIONS:
Procedure: Oral Glucose Tolerance Test (OGTT) — Subjects will have glucose administered enterally and blood will be drawn to measure its kinetics.
  Other Names: OGTT
Drug: Human Ghrelin — Human ghrelin will be administered by IV at two of the four study visits in conjunction with the OGTT.
  Other Names: Ghrelin
Drug: Saline — Saline Infusion will be administered by IV at two of the four study visits in conjunction with the OGTT to serve as a placebo comparator for the human ghrelin infusions.
  Other Names: NaCl, sodium chloride

SUMMARY:
The purpose of this study is to determine if the altered nutrient exposure to the GI tract after bariatric surgery reveals a negative incretin effect of ghrelin.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2
* Age 21-65 years
* Weight ≤ 200 kg

Exclusion Criteria:

* Type 2 or Type 1 diabetes
* Medications that alter insulin sensitivity or carbohydrate metabolism
* Positive pregnancy test
* Known history of intestinal diseases including, but not limited to, inflammatory bowel disease (e.g. Chronic Ulcerative Colitis, Crohn's disease, celiac sprue)
* Prior gastric or intestinal surgery or pancreas resection
* History of cardiovascular disease, including but not limited to: myocardial infarction, angioplasty, arrhythmia, uncontrolled hypertension
* History of chronic kidney disease or renal insufficiency; creatinine > 1.8 mg/dl.
* History of chronic liver disease, including but not limited to: cirrhosis, hepatitis, portal hypertension; AST and/or ALT > 2x the upper limit of normal.
* Abnormal ECG

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-08-21 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose levels with ghrelin versus saline. | 1 month (before and after surgery)
  The objective for this protocol is to determine if ghrelin infusion worsens glucose tolerance during jejunal administration of glucose and if the response is difference after bariatric surgery (RYGB or VSG).

SECONDARY OUTCOMES:
Plasma insulin levels | 1 month (before and after surgery)

OTHER OUTCOMES:
Plasma Levels of GLP-1 | 1 month (before and after surgery)
  Metabolic panel to include plasma levels of GLP-1
Plasma Levels of GIP | 1 month (before and after surgery)
  Metabolic panel to include plasma levels of GIP
Plasma Levels of leptin | 1 month (before and after surgery)
  Metabolic panel to include plasma levels of leptin
Plasma Levels of pancreatic polypeptide | 1 month (before and after surgery)
  Metabolic panel to include plasma levels of pancreatic polypeptide
Plasma Levels of Peptide YY (PYY) | 1 month (before and after surgery)
  Metabolic panel to include plasma levels of PYY
Plasma Levels of C-Peptide | 1 month (before and after surgery)
  Metabolic panel to include plasma levels of C-Peptide
Plasma Levels of glucagon | 1 month (before and after surgery)
  Metabolic panel to include plasma levels of glucagon
Plasma Levels of Cholecystokinin (CCK) | 1 month (before and after surgery)
Plasma Levels of Cholecystokinin Adrenocorticotropic Hormone (ACTH) | 1 month (before and after surgery)
Plasma Levels of Human Growth Hormone (HGH) | 1 month (before and after surgery)
Plasma Levels of Cortisol | 1 month (before and after surgery)
Plasma Levels of insulin-like growth factor 1 (IGF-1) | 1 month (before and after surgery)
Acyl and desacyl ghrelin | 1 month (before and after surgery)
Plasma Levels of Bile Acids | 1 month (before and after surgery)
Plasma Levels of Free Fatty Acids (FFAs) | 1 month (before and after surgery)
Plasma Levels of Triglycerides (TG) | 1 month (before and after surgery)
Performance on Visual Analog Scale for Hunger | 1 month (before and after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided